CLINICAL TRIAL: NCT06228573
Title: Combining Transcranial Direct Current Stimulation and Yoga for Improved Pain Management for Knee Osteoarthritis: A Pilot and Feasibility Trial
Brief Title: Transcranial Direct Current Stimulation and Yoga for Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Arthritis Society, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-0000000177
Record Dates: First submitted 2024-01-16; First posted 2024-01-29 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Yoga

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Active tDCS Arm:
  In Week 1, participants in the Active tDCS arm will undergo five in-person visits for the administration of active transcranial Direct Current Stimulation (tDCS). Subsequently, from Weeks 2 to 9, participants will receive weekly active tDCS sessions preceding the scheduled yoga sessions.
  For the active tDCS sessions, a constant current stimulator will be employed to deliver direct current through a pair of surface sponge electrodes (5×7 cm) soaked in saline. Participants will undergo anodal stimulation targeting the primary motor cortex (M1) contralateral to the most painful site (C3 or C4 based on the electroencephalogram 10/20 system). The cathodal electrode will be positioned on the supraorbital area contralateral to the anode. During active tDCS, a constant anodal current of 2 mA will be administered for 20 minutes, a duration known to enhance cortical excitability and alleviate pain. T
  Interventions: Procedure: Yoga
- Sham tDCS (Sham Comparator): Sham tDCS Arm:
  tDCS: In Week 1, participants in the Sham tDCS arm will attend five in-person visits for the administration of sham transcranial Direct Current Stimulation (tDCS). From Weeks 2 to 9, participants will receive weekly sham tDCS sessions before the scheduled yoga sessions.
  Constant current stimulator will be used to deliver direct current through a pair of surface sponge electrodes (5×7 cm) soaked in saline. Participants will undergo sham stimulation targeting the primary motor cortex (M1) contralateral to the most painful site (C3 or C4 based on the electroencephalogram 10/20 system).
  During sham tDCS, the electrodes will be placed in the same montage as the active tDCS; however, current will only be applied for the initial and final 30 seconds of the 20-minute session. Consequently, participants will experience the sensation of current ramping up and down but will receive no current for the remaining stimulation period.
  Interventions: Procedure: Yoga

INTERVENTIONS:
Procedure: Yoga — Yoga program: In weeks 2-9, participants will attend twice weekly 1-hour sessions of yoga led by a certified yoga instructor trained in the intervention by collaborator Pearson. Videos will be provided for completion of home sessions. The yoga program is based on the Pain Care Aware certification program.38 Details of the program as well as the training of instructors are provided in the appendices. Briefly, classes will consist of 3 parts: centring and warming up aimed at regulating physiology prior to beginning the yoga postures; yoga postures and guided relaxation.

SUMMARY:
People with knee arthritis often experience constant pain, and current treatments aren't very effective. This can lead to limited movement and more health problems. Knee arthritis is a big part of healthcare costs in Canada, and its pain is a major reason people see doctors. The pain is linked to complex nervous system changes, making current treatments, like exercise, not very successful.

To address this, researchers suggest a new approach combining two things: a brain stimulation technique called Transcranial Direct Current Stimulation (tDCS) and yoga. TDCS helps with pain by changing how the brain works, and yoga, a safe practice, focuses on overall well-being. Together, the investigators aim to improve how the nervous system works from top to bottom.

The research project wants to change how the arthritis pain is being managed by focusing on how it works. The investigators plan to test this combo in a study comparing real tDCS plus yoga with fake tDCS plus yoga. The investigators will look not only at pain but also at other measures related to pain and how the nervous system works. This new mix could be a meaningful way to reduce pain for people with knee arthritis.

DETAILED DESCRIPTION:
Background:

'Omnipresent' is a common word that people living with knee osteoarthritis (KOA) use to describe the associated pain, with its unpredictability causing physical, social and emotional disruption. For many, KOA pain leads to limited mobility, reduced quality of life and increased healthcare costs KOA pain and its mechanisms are known to be complex, with alterations in nervous system signaling (ANSS) leading to persistent pain, and treatment failure to guideline-based care. Unfortunately, there is a lack of effective conservative treatments for KOA pain, including exercise which elicits only modest analgesic effects and has little impact on ANSS. To improve conservative pain management for people with KOA, it is imperative to design mechanism informed interventions and explore bold new ways to modulate ANSS to optimize patient outcomes.

The investigators' novel intervention is focused on addressing the biomarker of ANSS. The investigators' solution involves using non-invasive brain stimulation (NIBS) in the form of transcranial direct current stimulation (tDCS), paired with the mind-body practice of yoga, to modify neural pathways. This is a promising and safe alternative to medications - which risk habituation, adverse events, and addiction - and that builds on the limited efficacy of performing/examining exercise in isolation. To the investigators' knowledge, this is the first trial to use this combination for chronic pain and in people with KOA. The investigators have chosen this combination as tDCS has the potential to produce synergistic nervous system effects with yoga and bolster impacts on pain.

tDCS alleviates pain in older adults with KOA, particularly when combined with strengthening exercise or mindfulness. tDCS has demonstrated improved efficiency of conditioned pain modulation (CPM) resulting in pain reduction in older adults with KOA displaying deficient CPM. Meta-analyses of tDCS for the treatment of chronic pain report small to moderate effects on pain reduction, while a meta-analysis of NIBS (including tDCS) plus exercise showed moderate to large effect sizes (-0.62) compared to sham NIBS plus exercise.

The investigators' approach combining 13 sessions of tDCS with yoga provides the benefits of strengthening and mindfulness in addition to nervous system regulation with the potential to produce large effects for pain reduction.

Yoga modulates brain networks and is safe and accessible for many with KOA Importantly, yoga is safe for people with comorbidities through its combination of physical postures, breathing exercises, meditation and relaxation that are hypothesized to reduce pain by regulating top down and bottom-up input into the physiological systems modulating nociceptive signals. Evidence from fMRI studies indicates that yoga modifies functional connectivity in networks involved in chronic pain. Yoga is conditionally recommended by KOA guidelines due to low quality evidence and few studies.

The current project seeks to shift the current paradigm for conservative pain management for people with KOA by assessing a pain mechanism informed treatment strategy in a multi-center pilot and feasibility randomized controlled trial. The investigators hypothesize that real tDCS and yoga will provide clinically meaningful reductions in pain compared to sham tDCS and yoga.

This is a feasibility and pilot double-blind, randomized sham-controlled multi-center, two-arm clinical trial with a 1:1 allocation ratio. Participants will be randomized to receive active or sham tDCS and yoga for 9 weeks. Follow-up will occur at the end of the intervention and at 3 months. The Conceptual Framework for Defining Feasibility and Pilot studies, and the Standard Protocol Items- Recommendations for Intervention Trials will be used. Study results will be reported using the extended CONSORT guideline for pilot trials and the Check List Standardizing the Reporting of Interventions For Yoga (CLARIFY).

ELIGIBILITY:
Inclusion Criteria:

* community dwelling adults from Sherbrooke, Quebec, Hamilton and London, Ontario fulfilling the NICE criteria for KOA
* ≥45 years of age
* Diagnosis of Knee osteoarthritis OR
* Having movement-related joint pain with either no morning knee stiffness or stiffness of 30 minutes or less AND
* Experiencing an average pain intensity of ≥3 /10 in the past month

Exclusion Criteria:

* Systemic inflammatory arthritis.
* Any knee injection in the past 3 months.
* Inability to independently get up and down from the floor.
* Lower limb trauma or surgery within the last 6 months.
* Current participation in another OA clinical trial.
* Use of mobility aids.
* Currently receiving care for KOA pain (e.g., physiotherapy).
* Planned absences exceeding 1 week.
* Contraindications to transcranial direct current stimulation (tDCS) such as neurological or neuropsychiatric conditions.
* History of brain surgery or tumor.
* Metallic implants.
* Epilepsy or history of substance abuse or dependence.
* Cochlear or ocular implant.
* Presence of a pacemaker or cardiac defibrillator.
* Eczema on the scalp.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of complete follow up | 9 weeks and 3 months
  Percentage rate measured by those at baseline completing study follow up measures

SECONDARY OUTCOMES:
Brief Pain Inventory - Numeric Rating Scale | 9 weeks and 3 months
  The BPI uses 4 questions to ask about worst and least pain intensity in the past 24 hours, pain on average and pain right now. Questions are rated on an 11-point scale where patients select a rating between 0-10 with zero representing 'no pain' and 10 representing the 'worst imaginable pain'. The Numeric Rating Scale is reported to have excellent inter-rater reliability and acceptable validity in people with KOA.
Modified Charlson Comorbidity Index (CCI) | 9 weeks and 3 months
  To assesses the presence of 19 comorbidities in participants. The CCI has been used in many patient populations including knee osteoarthritis
Endogenous pain modulation | 9 weeks
  CPM will be assessed in the following steps: 1) at the anterior shin on the unaffected knee, an ascending measure of pressure pain threshold (PPT) will be evaluated, inducing a pain rating of 3/10. 2) At the opposite volar forearm, a conditioning stimulus in the form of forearm ischemia using a blood pressure cuff and squeezing a stress ball until a pain rating of 5/10 is reached, 3) PPT at the anterior shin will be repeated with the cuff remaining inflated2, 4) an index will be created by calculating the percent efficiency of CPM (%CPM) as PPT2/PPT1, multiplied by 100; whereby %CPM ≤ 100 indicates inefficient pain modulation. CPM testing has demonstrated good intra-session reliability.
Pain interference | 9 weeks and 3 months
  The Brief Pain Inventory5 assesses pain interference through 7 items general activity, mood, walking, normal work, relations with others, sleeping, enjoyment of life rated from 0 (does not interfere) to 10 (completely interferes).
Pain catastrophizing | 9 weeks and 3 months
  Pain Catastrophizing Scale (PCS); The PCS is a 13-item self-reporting instrument for catastrophizing in the context of actual or anticipated pain, with higher scores indicating higher pain catastrophizing. The validity of the PCS for measuring pain catastrophizing in people with KOA has been reported.
Hospital Anxiety and Depression Scale (HADS) | 9 weeks and 3 months
  The HADS is a brief and reliable measure of emotional distress in general in chronic populations. Validity and reliability of the HADS have been previously established. Higher scores on the HADS indicate increased severity of anxiety and depression symptoms.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 9 weeks and 3 months
  The KOOS pain and function in daily living and QoL subscales will be used to assess self-reported opinions about patients' knee and associated problems. Scores range from 0-100 with zero representing extreme knee problems and 100 representing no knee problems. KOOS has adequate internal consistency and validity in people with KOA.
Multi-joint pain; Body diagram | 9 weeks and 3 months
  Participants will be asked to indicate any other areas where they experience pain (e.g., neck, shoulders, back) on a body diagram which will be summed to form a count. Body diagrams are a reliable method for indication of painful body parts.
Knee Awareness | 9 weeks and 3 months
  Fremantle knee awareness questionnaire; Developed from the low back version, the scale has good reliability and is correlated with pain in motion, disability, catastrophizing, fear of movement, and anxiety. It consists of 9 items rated from never to always. Higher scores indicate lower knee awareness.
Functional leg strength | 9 weeks
  Stair climb test; The OARSI recommended test will measure the time (in seconds) it takes to ascend and descend a flight of stairs consisting of 9 steps and a handrail. The test has excellent reliability and responsiveness.
Medication use | 9 weeks and 3 months
  Survey question; Participants will be asked to indicate use of any SSRI or SNRI medication that they take regularly and which can impact neuromodulation. Use of these medications will be adjusted for in our model
Adverse events | 9 weeks
  Survey question; We will monitor adverse events related to tDCS using the following questionnaire: Do you experience any of the following symptoms or side-effects? Headache Neck pain Scalp pain Tingling Itching Burning sensation Skin redness Sleepiness Trouble concentrating Acute mood change Others (specify) rated as absent, mild, moderate or severe and then If present: Is this related to tDCS? (1, none ; 2, remote; 3, possible; 4, probable; 5, definite).
  We will also monitor adverse events related to yoga by asking the participants to report any problems that they experience after the yoga class that last for more than two days and/or urged them to seek treatment or if they experience any adverse events during the class (such as falls or injuries)
Patient global impression of change | 9 weeks and 3 months
  At the end of the program, participants will be asked to rate the amount of change on a 7 point scale experienced ranging from very much improved to very much worse. The scale is widely used and validated as a measure of minimally important change
Blinding effectiveness | 3 months
  Participants will be asked to indicate which intervention group they believed they were in.
Usefulness of the program for managing knee OA measured on a 5 point Likert scale | 9 weeks
  Likert scale anchored from Not useful at all to very useful
Frequency of the program measured on a 5 point Likert scale | 9 weeks
  Likert scale anchored from not frequent enough to Frequent enough
Duration of the program on a 5 point Likert scale | 9 weeks
  Likert scale anchored from not long enough to long enough
Acceptability of the delivery of the brain stimulation on a 5 point Likert scale | 9 weeks
  Likert scale anchored from not at all accepted to very acceptable
Acceptability of the delivery of the yoga session of the program on a 5 point Likert scale | 9 weeks
  Likert scale anchored from not at all accepted to very acceptable
How likely are you to recommend the program you attended for others with knee OA? | 9 weeks
  Likert scale anchored from not at all likely to very likely
How burdensome did you find completing the questionnaires? | 3 months
  10 point scale- burdensomeness rating between 0 (no burden at all) to 10 (very much a burden)
How burdensome did you find completing the physical assessments? | 9 weeks
  10 point scale- burdensomeness rating between 0 (no burden at all) to 10 (very much a burden)
rate of adherence measured by percentage of sessions attended and home sessions completed | 9 weeks
  adherence rate calculated from attendance and exercise tracking sheets

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carlesso, PhD, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - University of Western Ontario, London, Ontario
  - Université de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallis JA, Taylor NF, Bunzli S, Shields N. Experience of living with knee osteoarthritis: a systematic review of qualitative studies. BMJ Open. 2019 Sep 24;9(9):e030060. doi: 10.1136/bmjopen-2019-030060. PMID 31551381
- [Background] Calders P, Van Ginckel A. Presence of comorbidities and prognosis of clinical symptoms in knee and/or hip osteoarthritis: A systematic review and meta-analysis. Semin Arthritis Rheum. 2018 Jun;47(6):805-813. doi: 10.1016/j.semarthrit.2017.10.016. Epub 2017 Oct 31. PMID 29157670
- [Background] Kendzerska T, Juni P, King LK, Croxford R, Stanaitis I, Hawker GA. The longitudinal relationship between hand, hip and knee osteoarthritis and cardiovascular events: a population-based cohort study. Osteoarthritis Cartilage. 2017 Nov;25(11):1771-1780. doi: 10.1016/j.joca.2017.07.024. Epub 2017 Aug 9. PMID 28801210
- [Background] Arthritis Alliance of Canada. The Impact of Arthritis in Canada: Today and over the Next 30 years. Executive Summary. 2011.
- [Background] Sharif B, Kopec JA, Wong H, Anis AH. Distribution and Drivers of Average Direct Cost of Osteoarthritis in Canada From 2003 to 2010. Arthritis Care Res (Hoboken). 2017 Feb;69(2):243-251. doi: 10.1002/acr.22933. PMID 27159532
- [Background] Neogi T. The epidemiology and impact of pain in osteoarthritis. Osteoarthritis Cartilage. 2013 Sep;21(9):1145-53. doi: 10.1016/j.joca.2013.03.018. PMID 23973124
- [Background] Fingleton C, Smart K, Moloney N, Fullen BM, Doody C. Pain sensitization in people with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Jul;23(7):1043-56. doi: 10.1016/j.joca.2015.02.163. Epub 2015 Mar 5. PMID 25749012
- [Background] Carlesso LC, Segal NA, Frey-Law L, Zhang Y, Na L, Nevitt M, Lewis CE, Neogi T. Pain Susceptibility Phenotypes in Those Free of Knee Pain With or at Risk of Knee Osteoarthritis: The Multicenter Osteoarthritis Study. Arthritis Rheumatol. 2019 Apr;71(4):542-549. doi: 10.1002/art.40752. Epub 2019 Feb 7. PMID 30307131
- [Background] O'Leary H, Smart KM, Moloney NA, Blake C, Doody CM. Pain sensitization associated with nonresponse after physiotherapy in people with knee osteoarthritis. Pain. 2018 Sep;159(9):1877-1886. doi: 10.1097/j.pain.0000000000001288. PMID 29794610
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] Fernandes L, Hagen KB, Bijlsma JW, Andreassen O, Christensen P, Conaghan PG, Doherty M, Geenen R, Hammond A, Kjeken I, Lohmander LS, Lund H, Mallen CD, Nava T, Oliver S, Pavelka K, Pitsillidou I, da Silva JA, de la Torre J, Zanoli G, Vliet Vlieland TP; European League Against Rheumatism (EULAR). EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis. Ann Rheum Dis. 2013 Jul;72(7):1125-35. doi: 10.1136/annrheumdis-2012-202745. Epub 2013 Apr 17. PMID 23595142
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Hall M, Dobson F, Plinsinga M, Mailloux C, Starkey S, Smits E, Hodges P, Vicenzino B, Schabrun SM, Masse-Alarie H. Effect of exercise on pain processing and motor output in people with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2020 Dec;28(12):1501-1513. doi: 10.1016/j.joca.2020.07.009. Epub 2020 Aug 9. PMID 32783909
- [Background] Ahn H, Sorkpor S, Miao H, Zhong C, Jorge R, Park L, Abdi S, Cho RY. Home-based self-administered transcranial direct current stimulation in older adults with knee osteoarthritis pain: An open-label study. J Clin Neurosci. 2019 Aug;66:61-65. doi: 10.1016/j.jocn.2019.05.023. Epub 2019 May 29. PMID 31153751
- [Background] Ahn H, Suchting R, Woods AJ, Miao H, Green C, Cho RY, Choi E, Fillingim RB. Bayesian analysis of the effect of transcranial direct current stimulation on experimental pain sensitivity in older adults with knee osteoarthritis: randomized sham-controlled pilot clinical study. J Pain Res. 2018 Sep 27;11:2071-2082. doi: 10.2147/JPR.S173080. eCollection 2018. PMID 30310309
- [Background] Tavares DRB, Okazaki JEF, Santana MVA, Pinto ACPN, Tutiya KK, Gazoni FM, Pinto CB, Santos FC, Fregni F, Trevisani VFM. Motor cortex transcranial direct current stimulation effects on knee osteoarthritis pain in elderly subjects with dysfunctional descending pain inhibitory system: A randomized controlled trial. Brain Stimul. 2021 May-Jun;14(3):477-487. doi: 10.1016/j.brs.2021.02.018. Epub 2021 Mar 5. PMID 33684598
- [Background] Pinto CB, Teixeira Costa B, Duarte D, Fregni F. Transcranial Direct Current Stimulation as a Therapeutic Tool for Chronic Pain. J ECT. 2018 Sep;34(3):e36-e50. doi: 10.1097/YCT.0000000000000518. PMID 29952860
- [Background] Lee PG, Jackson EA, Richardson CR. Exercise Prescriptions in Older Adults. Am Fam Physician. 2017 Apr 1;95(7):425-432. PMID 28409595
- [Background] Solomon DH, Schneeweiss S, Glynn RJ, Kiyota Y, Levin R, Mogun H, Avorn J. Relationship between selective cyclooxygenase-2 inhibitors and acute myocardial infarction in older adults. Circulation. 2004 May 4;109(17):2068-73. doi: 10.1161/01.CIR.0000127578.21885.3E. Epub 2004 Apr 19. PMID 15096449
- [Background] Pearson N, Prosko S, Sullivan M, Taylor MJ. White Paper: Yoga Therapy and Pain-How Yoga Therapy Serves in Comprehensive Integrative Pain Management, and How It Can Do More. Int J Yoga Therap. 2020 Jan 1;30(1):117-133. doi: 10.17761/2020-D-19-00074. PMID 32412808
- [Background] MacKay C, Jaglal SB, Sale J, Badley EM, Davis AM. A qualitative study of the consequences of knee symptoms: 'It's like you're an athlete and you go to a couch potato'. BMJ Open. 2014 Oct 16;4(10):e006006. doi: 10.1136/bmjopen-2014-006006. PMID 25324325
- [Background] Nyvang J, Hedstrom M, Gleissman SA. It's not just a knee, but a whole life: A qualitative descriptive study on patients' experiences of living with knee osteoarthritis and their expectations for knee arthroplasty. Int J Qual Stud Health Well-being. 2016 Mar 31;11:30193. doi: 10.3402/qhw.v11.30193. eCollection 2016. PMID 27036130
- [Background] Chang WJ, Bennell KL, Hodges PW, Hinman RS, Young CL, Buscemi V, Liston MB, Schabrun SM. Addition of transcranial direct current stimulation to quadriceps strengthening exercise in knee osteoarthritis: A pilot randomised controlled trial. PLoS One. 2017 Jun 30;12(6):e0180328. doi: 10.1371/journal.pone.0180328. eCollection 2017. PMID 28665989
- [Background] Ahn H, Zhong C, Miao H, Chaoul A, Park L, Yen IH, Vila MA, Sorkpor S, Abdi S. Efficacy of combining home-based transcranial direct current stimulation with mindfulness-based meditation for pain in older adults with knee osteoarthritis: A randomized controlled pilot study. J Clin Neurosci. 2019 Dec;70:140-145. doi: 10.1016/j.jocn.2019.08.047. Epub 2019 Aug 14. PMID 31421990
- [Background] Cardenas-Rojas A, Pacheco-Barrios K, Giannoni-Luza S, Rivera-Torrejon O, Fregni F. Noninvasive brain stimulation combined with exercise in chronic pain: a systematic review and meta-analysis. Expert Rev Neurother. 2020 Apr;20(4):401-412. doi: 10.1080/14737175.2020.1738927. Epub 2020 Mar 14. PMID 32130037
- [Background] Sefat O, Salehinejad MA, Danilewitz M, Shalbaf R, Vila-Rodriguez F. Combined Yoga and Transcranial Direct Current Stimulation Increase Functional Connectivity and Synchronization in the Frontal Areas. Brain Topogr. 2022 Mar;35(2):207-218. doi: 10.1007/s10548-022-00887-z. Epub 2022 Jan 29. PMID 35092544
- [Background] Lauche R, Hunter DJ, Adams J, Cramer H. Yoga for Osteoarthritis: a Systematic Review and Meta-analysis. Curr Rheumatol Rep. 2019 Jul 23;21(9):47. doi: 10.1007/s11926-019-0846-5. PMID 31338685
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Moonaz S, Nault D, Cramer H, Ward L. CLARIFY 2021: explanation and elaboration of the Delphi-based guidelines for the reporting of yoga research. BMJ Open. 2021 Aug 5;11(8):e045812. doi: 10.1136/bmjopen-2020-045812. PMID 34353794
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Roizenblatt S, Fregni F, Gimenez R, Wetzel T, Rigonatti SP, Tufik S, Boggio PS, Valle AC. Site-specific effects of transcranial direct current stimulation on sleep and pain in fibromyalgia: a randomized, sham-controlled study. Pain Pract. 2007 Dec;7(4):297-306. doi: 10.1111/j.1533-2500.2007.00152.x. Epub 2007 Nov 6. PMID 17986164
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Kim YJ, Ku J, Kim HJ, Im DJ, Lee HS, Han KA, Kang YJ. Randomized, sham controlled trial of transcranial direct current stimulation for painful diabetic polyneuropathy. Ann Rehabil Med. 2013 Dec;37(6):766-76. doi: 10.5535/arm.2013.37.6.766. Epub 2013 Dec 23. PMID 24466511
- [Background] Mori F, Codeca C, Kusayanagi H, Monteleone F, Buttari F, Fiore S, Bernardi G, Koch G, Centonze D. Effects of anodal transcranial direct current stimulation on chronic neuropathic pain in patients with multiple sclerosis. J Pain. 2010 May;11(5):436-42. doi: 10.1016/j.jpain.2009.08.011. Epub 2009 Dec 16. PMID 20018567
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Kessler SK, Turkeltaub PE, Benson JG, Hamilton RH. Differences in the experience of active and sham transcranial direct current stimulation. Brain Stimul. 2012 Apr;5(2):155-62. doi: 10.1016/j.brs.2011.02.007. Epub 2011 Mar 27. PMID 22037128
- [Background] Palm U, Reisinger E, Keeser D, Kuo MF, Pogarell O, Leicht G, Mulert C, Nitsche MA, Padberg F. Evaluation of sham transcranial direct current stimulation for randomized, placebo-controlled clinical trials. Brain Stimul. 2013 Jul;6(4):690-5. doi: 10.1016/j.brs.2013.01.005. Epub 2013 Feb 8. PMID 23415938